CLINICAL TRIAL: NCT01368822
Title: Effect of Obesity on Long-term Clinical Outcomes After Kidney Donation
Acronym: R-21
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK078702-02
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Renal Dysfunction; Hypertension
MeSH Terms: conditions — Renal Insufficiency; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Several studies have shown that renal function in patients who have donated a kidney (but are otherwise healthy) remains stable and within normal limits. However, it is unclear how donor nephrectomy affects patient subsets with comorbidities, an issue that becomes relevant in the current environment where inclusion criteria are continuously becoming less stringent and more patients are being considered as potential donors.

In the present study, the investigators plan to evaluate long-term renal function in obese patients who have donated a kidney as part of a living donor renal transplant procedure. The investigators have selected this group because it is at higher risk for developing obesity-related complications such as diabetes and hypertension that may impair renal function, it is rapidly becoming a major subgroup in the kidney donor population, and no studies have systematically followed obese patients after kidney donation. Establishment of an appropriate control group is of primary importance in studies examining long-term outcomes. The investigators will also evaluate a 2-kidney control group to allow us to compare the individual and interactive effects of obesity and kidney donation on long-term renal function. Study participants will complete a medical questionnaire, undergo blood pressure measurements, and provide blood and urine samples for analysis of various metabolic parameters. Some study participants will have ambulatory blood pressure monitoring performed which involves application of an automated blood pressure cuff for 24 hours. Some study participants will also undergo direct measurements of glomerular filtration rate (GFR) with iohexol.

In the proposed research, the investigators hypothesize that obesity in kidney donors increases the likelihood of developing renal dysfunction and risk factors for cardiovascular disease (CVD) and may increase the likelihood even more than in healthy controls.

DETAILED DESCRIPTION:
In order to meet the growing demand for living donor kidneys, the inclusion criteria for prospective donors have become less selective, allowing previously ineligible patients to donate kidneys. One donor group that has become increasingly more utilized is the overweight patient. There is substantial evidence that overweight individuals are more susceptible to the development of renal disease either as a direct result of their weight or as a consequence of their obesity-related co-morbidities such as diabetes and hypertension. In addition, it appears that even mild renal dysfunction can increase the risk of developing CVD, which is already more common in this population. Despite these findings, very little is known about the individual and interactive effects of obesity and donation on the overall health of kidney donors. Our study addresses some of these questions by examining the effects of obesity on long-term renal function and development of cardiovascular risk factors such as hypertension, dyslipidemia, and metabolic syndrome in patients who donated a kidney at the University of California, San Francisco (UCSF) more than 5 years ago (1967-2006). The control group will comprise of all potential kidney donors at UCSF during this period who passed an initial medical screening evaluation but did not donate because they were found to be ABO- or crossmatch incompatible. The investigators believe that the results of the proposed study will be important in developing more precise guidelines for the selection and long-term health care maintenance of kidney donors.maintenance at all.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone donor nephrectomy as part of living donor kidney transplantation at UCSF between 1967 and 2006 (study patients).
* Patients who were accepted for kidney donation at UCSF between 1967 and 2006 but were excluded from donation due to blood type or crossmatch incompatibility with the recipient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients who underwent donor nephrectomy at UCSF more than 5 years ago and a 2-kidney control group which consist of prospective donors evaluated at UCSF who were found to be eligible for donation on the basis of a medical screening evaluation, but then were excluded due to ABO-incompatibility or positive crossmatch with the recipient.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States